CLINICAL TRIAL: NCT03146299
Title: Comparison of Total Laparoscopic Hysterectomy and Laparoscopic Assisted Vaginal Hysterectomy With Over Giant Uterus of Than 500g: A Randomized Controlled Trial
Brief Title: Comparison of TLH and LAVH With Over Than 500g
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Joong Sub Choi, Professor and Director of the Division of Gynecologic Oncology and Gynecologic Minimally Invasive Surgery, Full-time faculty of the Department of Obstetrics and Gynecology, Hanyang University College of Medicine, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYGY 4004
Record Dates: First submitted 2017-05-06; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Hysterectomy, Benign Uterine Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: TLH (Active Comparator)
  Interventions: Procedure: TLH vs LAVH
- Group B: LAVH (Active Comparator)
  Interventions: Procedure: TLH vs LAVH

INTERVENTIONS:
Procedure: TLH vs LAVH — TLH: The subjects undergoing laparoscopic hysterectomy with a giant uterus of 500 g or more
  LAVH: The subjects undergoing Laparoscopic Assisted Vaginal Hysterectomy with a giant uterus of 500 g or more
  Other Names: TLH: Total Laparoscopic Hysterectomy, LAVH: Laparoscopic Assisted Vaginal Hysterectomy

SUMMARY:
Since the introduction of total laparoscopic hysterectomy in 1989, laparoscopic gynecologic surgery has undergone many advances. TLH or LAVH has the advantages of faster recovery, fewer complications and shorter hospitalization compared to total abdominal hysterectomy.

However, the hysterectomy for giant uterus has the difficulty of delivering the uterus out of the body. According to the results of TLH, LAVH and abdominal hysterectomy, TLH and LAVH show the postoperative complications were less frequent (3) and the postoperative recovery (4) and return to daily life were faster than total abdominal hysterectomy (3) even if it took longer operation time.

Therefore, laparoscopic hysterectomy has many advantages over abdominal hysterectomy and indications are increasing. However, there has not yet been a direct comparison between TLH and VALH for large uterine surgery. In this study, we compared the results including the complications, hospitalization period and so on., in undergoing operation and post-operation between TLH and LAVH for the removal of giant uterus, which is predicted to be over 500 g.

ELIGIBILITY:
Inclusion Criteria:

* Have the indication for hysterectomy for a supposed benign uterine disease
* Have a giant uterus of 500g or more
* Estimation of uterine weight more than 500g
* Uterine myoma size at 4 months or more after pregnancy due to pelvic examination
* The length of the long axis of one uterine myoma is more than 8cm or the length of the long axis for over 2 uterine myomas is more than 6cm
* Have been not pregnant at the time of presentation
* Have been appropriated medical status for laparoscopic surgery (surgery (American Society of Anesthesiologists Physical Status classification 1 or 2)

Exclusion Criteria:

* Have a suspicion of malignancy or malignant tumors (cervical cancer, ovarian cancer, fallopian tube cancer, peritoneal cancer, Endometrial cancer)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 1 month after surgery
  Incidence of postoperative complications

REFERENCES:
- [Background] Dicker RC, Greenspan JR, Strauss LT, Cowart MR, Scally MJ, Peterson HB, DeStefano F, Rubin GL, Ory HW. Complications of abdominal and vaginal hysterectomy among women of reproductive age in the United States. The Collaborative Review of Sterilization. Am J Obstet Gynecol. 1982 Dec 1;144(7):841-8. doi: 10.1016/0002-9378(82)90362-3. PMID 7148906
- [Background] Carter JE, Ryoo J, Katz A. Laparoscopic-assisted vaginal hysterectomy: a case control comparative study with total abdominal hysterectomy. J Am Assoc Gynecol Laparosc. 1994 Feb;1(2):116-21. doi: 10.1016/s1074-3804(05)80773-x. PMID 9050472
- [Background] Hwang JL, Seow KM, Tsai YL, Huang LW, Hsieh BC, Lee C. Comparative study of vaginal, laparoscopically assisted vaginal and abdominal hysterectomies for uterine myoma larger than 6 cm in diameter or uterus weighing at least 450 g: a prospective randomized study. Acta Obstet Gynecol Scand. 2002 Dec;81(12):1132-8. doi: 10.1034/j.1600-0412.2002.811206.x. PMID 12519109